CLINICAL TRIAL: NCT06313476
Title: A Prospective, Observational Clinical Study of AMH Predicting Postchemotherapy Menopause in Premenopausal Breast Cancer Patients Who do Not Use OFS
Brief Title: AMH Predicts Postchemotherapy Menopause in Premenopausal Breast Cancer Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2024-030-01
Record Dates: First submitted 2024-03-05; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Premenopausal patients with early breast cancer who received chemotherapy (neoadjuvant chemotherapy or adjuvant chemotherapy) and did not use OFS ovarian suppression at the Breast Cancer Center of Sun Yat-sen Memorial Hospital, Sun Yat-sen University

SUMMARY:
To determine the accuracy of AMH postchemotherapy in predicting permanent menopause after chemotherapy in breast cancer patients who did not use OFS before menopause

DETAILED DESCRIPTION:
For early breast cancer women who are premenopausal, after receiving chemotherapy (neoadjuvant chemotherapy or adjuvant chemotherapy), not using OFS as ovarian suppression, AMH, E2 and FSH levels will be measured by blood sampling before chemotherapy, at the end of chemotherapy and 1 month, 3 months, 6 months, 12 months, 18 months and 24 months after chemotherapy. The menstrual status of patients will be also followed up. At several timing, investigators will analyze AMH level, E2 level, FSH level, proportion of unmeasured AMH (AMH≤0.02ng/ml), proportion of E2 that conforms to menopausal status (E2≤30ng/L), proportion of FSH that conforms to menopausal status (FSH > 30U/L), proportion of persistent amenia (no menstruation from the end of chemotherapy to the evaluation time) and incidence of adverse reactions

ELIGIBILITY:
Inclusion Criteria:

1. Age over 40(include 40 years old), or before 60, female
2. Primary invasive breast cancer diagnosed by histopathology, except of occult breast cancer, inflammatory breast cancer and Paget's disease
3. Operable patients with no distant metastases at diagnosis (stage T1-T3, any N, M0)
4. The patient was at premenopausal status when first diagnosed (had menstruation in the last 12 months or hormone levels not reached menopause when diagnosed, E2 > 30ng/L, FSH≤30U/L)
5. The patient has used chemotherapy (neoadjuvant chemotherapy or adjuvant chemotherapy) after diagnosis

Exclusion Criteria:

1. Age before 40, or over 60(include 60 years old)
2. Patient who accepted bilateral ovariectomy or ovarian radiotherapy
3. Patient who used gonadotropin-releasing hormone agonist ( GnRHa)
4. Stage IV (metastatic) breast cancer
5. The patient was at postmenopausal status when first diagnosed (no menstruation in the past 12 months or hormone levels reached menopause when diagnosed, E2≤30ng/L, FSH > 30U/L)
6. The patient has not used chemotherapy (neoadjuvant or adjuvant chemotherapy) since diagnosis
7. The investigator determines that the patient has any other condition that make her unfit to participate in the study

Ages: 40 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Premenopausal early breast cancer patients who do not use OFS as ovarian suppression after receiving chemotherapy (neoadjuvant chemotherapy or adjuvant chemotherapy) at the Breast Tumor Center of Sun Yat-sen Memorial Hospital, Sun Yat-sen University.
Sampling Method: Probability Sample
Enrollment: 153 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Anti-Mullerian Hormone | Before chemotherapy, within a week after last chemotherapy, 1,3,6,12,18,24 months after chemotherapy
  Blood Test

SECONDARY OUTCOMES:
Estradiol | Before chemotherapy, within a week after last chemotherapy, 1,3,6,12,18,24 months after chemotherapy
  Blood Test
Follicle Stimulating Hormone | Before chemotherapy, within a week after last chemotherapy, 1,3,6,12,18,24 months after chemotherapy
  Blood Test
Menstruation | Before chemotherapy, within a week after last chemotherapy, 1,3,6,12,18,24 months after chemotherapy
  Follow-up